CLINICAL TRIAL: NCT03836677
Title: A Randomized, Double-blind, Two Treatment, Two Period, Chronic Dosing (4 Weeks), Crossover, Multi-center Pilot Study to Evaluate the Effects of Budesonide/Glycopyrronium/Formoterol Fumarate and Glycopyrronium/Formoterol Fumarate on Specific Image Based Airway Volumes and Resistance in Subjects With Moderate to Severe COPD
Brief Title: A Study to Evaluate the Effects of BGF and GFF on Specific Image Based Airway Volumes and Resistance in Subjects With Moderate to Severe COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: D5980C00019
Record Dates: First submitted 2018-09-24; First posted 2019-02-11 (Actual); Results first posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BGF-GFF (Experimental): Subject first treated with Budesonide/Glycopyrronium/Formoterol Fumarate followed by a washout period then treated with Glycopyrronium/Formoterol Fumarate
  Interventions: Combination Product: BGF; Combination Product: GFF
- GFF-BGF (Experimental): Subject first treated with Glycopyrronium/Formoterol Fumarate followed by a washout period then treated with Budesonide/Glycopyrronium/Formoterol Fumarate
  Interventions: Combination Product: BGF; Combination Product: GFF

INTERVENTIONS:
Combination Product: BGF — Treatment with Budesonide/Glycopyrronium/FormoterolFumarate
Combination Product: GFF — Treatment with Glycopyrronium/Formoterol Fumarate

SUMMARY:
This is a randomised, controlled, two period cross-over, 4 weeks chronic dosing, study to evaluate the effects of Budesonide/Glycopyrronium/Formoterol Fumarate (BGF) and Glycopyrronium/Formoterol Fumarate (GFF) on airway dimensions.

DETAILED DESCRIPTION:
This is a randomised, controlled, two period cross-over, 4 weeks chronic dosing, study to evaluate the effects of Budesonide/Glycopyrronium/Formoterol Fumarate (BGF), and Glycopyrronium/Formoterol Fumarate (GFF), on specific image based airway volumes and resistance in subjects with moderate to severe Chronic Obstructive Pulmonary Disease. In this study, airway dimension parameters will be calculated for each of the active compounds.

This imaging methodology will allow an assessment of the extent of airway changes using a triple combination of Budesonide/Glycopyrronium/Formoterol Fumarate (BGF) and the dual combination Glycopyrronium/Formoterol Fumarate (GFF).

ELIGIBILITY:
Inclusion Criteria:

Subject must be 40 years to ≤80 years of age inclusive, at the time of signing the informed consent form at Visit 1.

* COPD Diagnosis: Subjects with an established clinical history of COPD
* Screening clinical laboratory tests must be acceptable to the Investigator.
* Screening ECG must be acceptable to the Investigator
* Individual Compliance: Subjects must be willing to remain at the study center as required per protocol to complete all visit assessments
* Patients should be on scheduled maintenance treatment with one or more inhaled bronchodilator therapies.

Exclusion Criteria:

* As judged by the investigator, any evidence of significant diseases other than COPD, i.e., disease or condition which, in the investigator's opinion makes it undesirable for the subject to participate in the trial.
* Spirometry Performance:

  1. Subjects who cannot perform acceptable spirometry, i.e., meet ATS/ERS acceptability criteria.
  2. Repeatability: Subjects who cannot perform technically acceptable spirometry in accordance with ATS repeatability criteria
* Cancer: Subjects who have cancer that has not been in complete remission for at least five years.
* Substance Abuse: Subjects, who in the opinion of the Investigator, significantly abuse alcohol or drugs
* Subjects who in the opinion of the investigator are unable to abstain from prohibited medications including LABA/LAMAs/ICS

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Research Site, Erpent, Belgium
- Netherlands (3):
  - Research Site, Eindhoven
  - Research Site, Groningen
  - Research Site, Zutphen

REFERENCES:
- [Derived] van den Berge M, De Backer J, Van Holsbeke C, De Backer W, Trivedi R, Jenkins M, Dorinsky P, Aurivillius M. Functional respiratory imaging assessment of budesonide/glycopyrrolate/formoterol fumarate and glycopyrrolate/formoterol fumarate metered dose inhalers in patients with COPD: the value of inhaled corticosteroids. Respir Res. 2021 Jul 1;22(1):191. doi: 10.1186/s12931-021-01772-2. PMID 34210340
- See also: Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5980C00019&attachmentIdentifier=a5d5dc54-7197-4031-9e83-0480baeaa3f2&fileName=d5980c00019-sap-ed-2_Redacted.pdf&versionIdentifier=
- See also: CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5980C00019&attachmentIdentifier=603a22eb-76ce-4e33-af2d-84d7b45e7bb8&fileName=d5980c00019-csp-v3_Redacted-v1.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study randomized 23 subjects at 4 study centers (1 center in Belgium and 3 centers in the Netherlands) from Feb 2019 to Nov 2019.
Pre-assignment Details: Subjects were randomized into 1 of 2 treatment sequences. Sequence 1 received BGF MDI in Period 1 followed by GFF MDI in Period 2. Sequence 2 received GFF MDI in Period 1 followed by BGF MDI in Period 2.
Groups:
- BGF MDI/GFF MDI: Budesonide/Glycopyrronium/Formoterol Fumarate Metered Dose Inhalation followed by Washout and then Glycopyrronium/Formoterol Fumarate Metered Dose Inhalation
- GFF MDI/BGF MDI: Glycopyrronium/Formoterol Fumarate Metered Dose Inhalation followed by Washout and then Budesonide/Glycopyrronium/Formoterol Metered Dose Inhalation
Period: Period 1
Arm/Group | BGF MDI/GFF MDI | GFF MDI/BGF MDI
Started | 13 | 10
Completed | 13 | 9
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Washout
Arm/Group | BGF MDI/GFF MDI | GFF MDI/BGF MDI
Started | 13 | 9
Completed | 13 | 9
Not Completed | 0 | 0
Period: Period 2
Arm/Group | BGF MDI/GFF MDI | GFF MDI/BGF MDI
Started | 13 | 9
Completed | 12 | 9
Not Completed | 1 | 0
Not completed — Severe non-compliance to protocol | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population - all subjects who were randomized to treatment.
Groups:
- Overall Study: ITT Population
Arm/Group | Overall Study
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] — ITT Population
  Years | 64.9 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants] — ITT Population
  Participants
    Female | 5
    Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants] — ITT Population
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 23
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Specific Image-based Airway Volume (siVaw)
Description: Specific image-based airway volume (SiVaw) measured in mL/L. Average across lobes, adjusted for lobe volume. Reported as ratio to baseline.
Time Frame: Baseline, Day 29
Population: ITT Population
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio to baseline
Groups:
- BGF MDI: Budesonide/Glycopyrronium/Formoterol Fumarate Metered Dose Inhalation
- GFF MDI: Glycopyrronium/Formoterol Fumarate Metered Dose Inhalation
Arm/Group | BGF MDI | GFF MDI
Number analyzed (Participants) | 20 | 21
Ratio to baseline | 1.72 [1.38 to 2.13] | 1.53 [1.28 to 1.83]
Statistical Analysis 1: Comparison: BGF MDI; Test type: Other; p < 0.0001, t-test, 2 sided — Statistical significance assessed using Hochberg's procedure applied across primary endpoints within each treatment; Within-group comparison to baseline using paired test; Geometric Mean ratio to baseline = 1.72, 95% CI 2-sided [1.38 to 2.13]
Statistical Analysis 2: Comparison: GFF MDI; Test type: Other; p < 0.0001, t-test, 2 sided — Statistical significance assessed using Hochberg's procedure applied across primary endpoints within each treatment; Within-group comparison to baseline using paired test; Geometric mean ratio to baseline = 1.53, 95% CI 2-sided [1.28 to 1.83]

2. Primary Outcome: Specific Image-based Airway Resistance (siRaw)
Description: Specific image-based airway resistance (siRaw) measured in kPa∙s. Average across lobes, adjusted for lobe volume. Reported as ratio to baseline.
Time Frame: Baseline, Day 29
Population: ITT Population
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio to baseline
Arm/Group | BGF MDI | GFF MDI
Number analyzed (Participants) | 20 | 21
Ratio to baseline | 0.50 [0.39 to 0.63] | 0.52 [0.40 to 0.67]
Statistical Analysis 1: Comparison: BGF MDI; Test type: Other; p < 0.0001, t-test, 2 sided — Statistical significance assessed using Hochberg's procedure applied across primary endpoints within each treatment; Within-group comparison to baseline using paired test; Geometric mean ratio to baseline = 0.50, 95% CI 2-sided [0.39 to 0.63]
Statistical Analysis 2: Comparison: GFF MDI; Test type: Other; p < 0.0001, t-test, 2 sided — Statistical significance assessed using Hochberg's procedure applied across primary endpoints within each treatment; Within-group comparison to baseline using paired test; Geometric mean ratio to baseline = 0.52, 95% CI 2-sided [0.40 to 0.67]

3. Secondary Outcome: Image-based Airway Volume (iVaw)
Description: Image-based Airway Volume (iVaw) measured in mL. Average across lobes, without adjustment for lobe volume. Reported as ratio to baseline.
Time Frame: Baseline, Day 29
Population: ITT Population
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio to baseline
Arm/Group | BGF MDI | GFF MDI
Number analyzed (Participants) | 20 | 21
Ratio to baseline | 1.70 [1.37 to 2.11] | 1.51 [1.26 to 1.80]
Statistical Analysis 1: Comparison: BGF MDI; Test type: Other; p < 0.0001, t-test, 2 sided; Within-group comparison to baseline using paired test; Geometric mean ratio to baseline = 1.70, 95% CI [1.37 to 2.11]
Statistical Analysis 2: Comparison: GFF MDI; Test type: Other; p = 0.0001, t-test, 2 sided; Within-group comparison to baseline using paired test; Geometric mean ratio to baseline = 1.51, 95% CI 2-sided [1.26 to 1.80]

4. Secondary Outcome: Image-based Airway Resistance (iRaw)
Description: Image-based airway resistance (iRaw) measured in kPa∙s/L. Average across lobes, without adjustment for lobe volume. Reported as ratio to baseline.
Time Frame: Baseline, 29 Days
Population: ITT Population
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio to baseline
Arm/Group | BGF MDI | GFF MDI
Number analyzed (Participants) | 20 | 21
Ratio to baseline | 0.50 [0.40 to 0.63] | 0.52 [0.40 to 0.68]
Statistical Analysis 1: Comparison: BGF MDI; Test type: Other; p < 0.0001, t-test, 2 sided; Within-group comparison to baseline using paired test; Geometric mean ratio to baseline = 0.50, 95% CI 2-sided [0.40 to 0.63]
Statistical Analysis 2: Comparison: GFF MDI; Test type: Other; p < 0.0001, t-test, 2 sided; Within-group comparison to baseline using paired test; Geometric mean ratio to baseline = 0.52, 95% CI 2-sided [0.40 to 0.68]

5. Secondary Outcome: Forced Expiratory Volume in One Second (Post-dose FEV1).
Description: Change from baseline in Forced Expiratory Volume in One Second (Post-dose FEV1).
Time Frame: Baseline 29 Days
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: L
Arm/Group | BGF MDI | GFF MDI
Number analyzed (Participants) | 21 | 21
L | 0.346 [0.182 to 0.509] | 0.273 [0.140 to 0.405]
Statistical Analysis 1: Comparison: BGF MDI; Test type: Other; p = 0.0003, t-test, 2 sided; Within-group comparison to baseline using paired test; Mean Change from Baseline = 0.346, 95% CI 2-sided [0.182 to 0.509]
Statistical Analysis 2: Comparison: GFF MDI; Test type: Other; p = 0.0004, t-test, 2 sided; Within-group comparison to baseline using paired test; Mean Change from Baseline = 0.273, 95% CI 2-sided [0.140 to 0.405]

6. Secondary Outcome: Functional Residual Capacity (FRC)
Description: Change from baseline in Functional residual capacity (FRC).
Time Frame: Baseline, Day 29
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: L
Arm/Group | BGF MDI | GFF MDI
Number analyzed (Participants) | 22 | 21
L | -0.28 [-0.77 to 0.21] | -0.50 [-0.81 to -0.18]
Statistical Analysis 1: Comparison: BGF MDI; Test type: Other; p = 0.2515, t-test, 2 sided; Within-group comparison to baseline using paired test; Mean ratio to baseline = -0.28, 95% CI 2-sided [-0.77 to 0.21]
Statistical Analysis 2: Comparison: GFF MDI; Test type: Other; p = 0.0040, t-test, 2 sided; Within-group comparison to baseline using paired test; Mean ratio to baseline = -0.50, 95% CI 2-sided [-0.81 to -0.18]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from visit 2 throughout the treatment period and including the follow-up period telephone call.
Description: The Safety Population was defined as all subjects who were randomized to treatment and received at least one dose of study treatment. Serious adverse events were collected visit 2 throughout the treatment period and including the follow-up period telephone call.
Groups:
- BGF MDI: Budoesonide/Glycopyrronium/Formoterol Fumarate Metered Dose Inhalation
Arm/Group | BGF MDI | GFF MDI
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 2/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGF MDI (N=22) | GFF MDI (N=23)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGF MDI (N=22) | GFF MDI (N=23)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-07-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT03836677/Prot_001.pdf
  • Statistical Analysis Plan (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT03836677/SAP_002.pdf